CLINICAL TRIAL: NCT04919538
Title: Longitudinal Study for Relapsing Polychondritis
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: VCRC5508
Record Dates: First submitted 2021-05-11; First posted 2021-06-09 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Relapsing Polychondritis; Vasculitis
Keywords: RP
MeSH Terms: conditions — Polychondritis, Relapsing; Vasculitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relapsing Polychondritis Cohort

SUMMARY:
Relapsing polychondritis (RP) is a rare systemic inflammatory disease characterized by recurrent inflammation of cartilage including ears, nose, tracheobronchial tree, chest wall and joints. Less commonly, it can cause inflammation of eyes, vasculature, nervous system, skin and inner ear. The purpose of this study is to study the pathogenesis of RP.

DETAILED DESCRIPTION:
Relapsing polychondritis (RP) is a rare systemic inflammatory disease characterized by recurrent inflammation of cartilage including ears, nose, tracheobronchial tree, chest wall and joints. Less commonly, it can cause inflammation of eyes, vasculature, nervous system, skin and inner ear. There is variability in organ-system involvement and the disease course is relapsing making the diagnosis challenging. Delay in diagnosis can lead to end-organ damage and significant morbidity and mortality. There are no biomarkers or blood tests that can assist with assignment of a diagnosis.

Development of this longitudinal cohort and multicenter approach offers the potential to generate new insights and generate new questions regarding the immunology of the disease. Attainment of a better understanding of the mechanisms and trajectory of inflammation may yield insights into potential new diagnostic and treatment strategies.

Study visits will occur every 6 months, or annually. Blood and urine collection will occur at every visit. A physical exam and medical and medication history will at every visit; also, participants will be asked to complete several questionnaires to assess disease activity, health status, and tobacco, alcohol, and drug use.

ELIGIBILITY:
Inclusion Criteria:

* 1. Any subject considered to have a diagnosis of relapsing polychondritis according to the investigator.

Exclusion Criteria:

* 1. Inability to provide consent, or in the case of minors, assent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with relapsing polychondritis (RP). Enrollment will be sequential and participants will have disease in various stages and of different duration.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the pathogenesis of relapsing polychondritis using disease history. | Study completion; from baseline through month 36.
  To study the manner of development of disease in patients affected with relapsing polychondritis.

SECONDARY OUTCOMES:
PROMIS Questionnaires | Baseline, month 6, month 12, month 18, month 24, month 30, month 36
  Questions will ask about fatigue on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 6, month 12, month 18, month 24, month 30, month 36
  Questions will ask about pain interference on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 6, month 12, month 18, month 24, month 30, month 36
  Questions will ask about physical function on the PROMIS short form.
PROMIS Questionnaires | Baseline, month 6, month 12, month 18, month 24, month 30, month 36
  Questions will ask about global health on the PROMIS short form.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Merkel, MD, MPH, Study Director — University of Pennsylvania; Shubhasree Banerjee, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Relapsing Polychondritis Foundation — https://polychondritis.org
- See also: Vasculitis Clinical Research Consortium — https://www.rarediseasesnetwork.org/vcrc
- See also: Rare Diseases Clinical Research Network (RDCR) — http://www.rarediseasesnetwork.org/